CLINICAL TRIAL: NCT01640444
Title: Randomized Phase II Study to Explore the Influence of BRAF and PIK3K Status on the Efficacy of FOLFIRI Plus Bevacizumab or Cetuximab, as First Line Therapy of Patients With RAS Wild-type Metastatic Colorectal Carcinoma and < 3 Circulating Tumor Cells
Brief Title: Influence of BRAF and PIK3K Status on the Efficacy of 5-Fluorouracil/Leucovorin/Oxaliplatin (FOLFIRI) Plus Bevacizumab or Cetuximab in Patients With RAS Wild-type Metastatic Colorectal Carcinoma and < 3 Circulating Tumor Cells (CTC)
Acronym: VISNU-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-12-02; 2012-000840-90 (EudraCT Number)
Record Dates: First submitted 2012-06-13; First posted 2012-07-13 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer Metastatic
Keywords: colorectal carcinoma; BRAF and PIK3K; FOLFIRI -Bevacizumab -Cetuximab; circulating tumor cells
MeSH Terms: conditions — Colorectal Neoplasms; Hereditary Sensory and Autonomic Neuropathies; Neoplastic Cells, Circulating | interventions — Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): FOLFIRI+bevacizumab
  Interventions: Drug: FOLFIRI + bevacizumab
- B (Experimental): FOLFIRI + cetuximab
  Interventions: Drug: FOLFIRI + cetuximab

INTERVENTIONS:
Drug: FOLFIRI + bevacizumab — * Bevacizumab 5 mg/kg iv, followed by
  * Irinotecan 180 mg/m2 iv administered over a period of 30-90 minutes, followed by
  * Leucovorin (LV) 400 mg/m2 iv administered over a period of 2 hours, followed by
  * 5-FU 400 mg/m2 iv bolus, followed by
  * 5-FU 2,400 mg/m2 for 46 h continuous infusion. This treatment will start on day 1 and will be repeated every 2 weeks (1 cycle).
  Arms: A
Drug: FOLFIRI + cetuximab — * Cetuximab in an initial 120-minute infusion on day 1 of 400 mg/m2, followed by 60-minute infusions of cetuximab at a dose of 250 mg/m2, once weekly
  * FOLFIRI:
    * Irinotecan 180 mg/m2 iv administered over a period of 30-90 minutes, followed by
    * Leucovorin (LV) 400 mg/m2 iv administered over a period of 2 hours, followed by
    * 5-FU 400 mg/m2 iv bolus, followed by
    * 5-FU 2,400 mg/m2 for 46 h continuous infusion FOLFIRI will be given after the cetuximab infusion on day 1 of each period (every 2 weeks: 1 cycle).
  Arms: B

SUMMARY:
The purpose of the study is to explore the influence of BRAF and PIK3K status on the efficacy of FOLFIRI plus Bevacizumab or Cetuximab, as first line therapy of patients with RAS wild-type metastatic colorectal carcinoma and < 3 circulating tumor cells

ELIGIBILITY:
Inclusion Criteria:

1. Patient's Informed consent in written.
2. Age between 18-70 years old.
3. ECOG 0-1.
4. Life expectancy of at least 3 months.
5. Histological confirmation of adenocarcinoma of the colon or rectum.
6. Sample of tumour tissue available for evaluation of genes RAS, BRAF and PI3K. To be included in the study patients should present < 3 CTC in peripheral blood and RAS wild-type present in the sample of tumor tissue.
7. Measurable metastatic stage IV disease with at least 1 measurable metastatic lesion following RECIST criteria v 1.1 (non suitable for radical surgery at the inclusion time).
8. Prior radiotherapy is allowed but must be completed at least 4 weeks before randomization (if applicable).
9. Adequate bone marrow, liver and renal function.
10. Women of childbearing potential must have a negative serum or urine pregnancy test. Postmenopausal women must have been amenorrheic for at least 12 months.Both men and women participating in this study must use adequate contraception.
11. Subject must have the ability, in the opinion of the investigator, to comply with all the study procedures and follow-up examinations.

Exclusion Criteria:

1. Previous chemotherapy for metastatic disease.
2. Prior treatment with Bevacizumab, or EGFR inhibitors
3. Any anticancer treatment (chemotherapy, hormonal treatment, radiation treatment, surgery , immunotherapy, biologic therapy or tumour embolization) within 4 weeks before randomization.
4. Use of any investigational drug within 4 weeks before start the treatment.
5. Clinical or radiographic evidence of brain metastasis.
6. Uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg on repeated measurement) despite optimal medical management.
7. Previous history of hypertensive encephalopathy or hypertensive crises.
8. Current or history of peripheral neuropathy > or equal to 1 NCICTCAE.
9. Patients classified as fragile according to criteria listed in the protocol.
10. Significant cardiovascular disease (e.g. AVC, myocardial infarction, within 6 months before randomization). Unstable angina, congestive heart failure New York Heart Association (NYHA) ≥ class II, arrhythmia that requires treatment within 3 months before randomization.
11. Significant vascular disease (e.g. aortic aneurism requiring surgical intervention, pulmonary embolic, peripheral arterial thrombosis) within 6 months before randomization.
12. Previous history of significant haemorrhage /severe, within 1 month before randomization.
13. Major surgery, open surgical biopsy or significant traumatic injury within 4 weeks before randomization.
14. Large bore needle biopsy of a major organ within 14 days before randomization. Placement of central venous access port > or equal to 7 days before randomization is permitted.
15. Evidence or history of bleeding diathesis or coagulopathy.
16. INR >1.5 within 14 days prior to starting study treatment. EXEMPTION: patients on full anticoagulation must have an in-range INR[usually between 2-3]. Any anticoagulation therapy must be at stable dosing prior to enrolment.
17. History of previous abdominal fistula or gastrointestinal perforation within 6 months before randomization.
18. Serious non-healing wound, ulcer or bone fracture.
19. Acute or sub-acute of intestinal occlusion or history of intestinal inflammatory disease.
20. History of uncontrolled convulsive crises.
21. History of pulmonary fibrosis, acute lung disease or interstitial pneumonia.
22. Chronic, actual o recent use (10 days prior first drug administration) of acetylsalicylic acic (aspirin) > 325 mg/day or clopidogrel (75mg/day) or other treatments that can cause gastrointestinal ulcer (low-dose aspirin is permitted < or equal to 325 mg/day).
23. Urinary protein excretion > or equal to 2+ (dipstick). If > or equal 2 g proteinuria is detected with dipstick, a 24-hour period urine test will be performed and the result should be < or equal to 1 g/24 hours to permit the inclusion of the patient in the clinical trial
24. Known human immunodeficiency virus infection or chronic hepatitis B or C infection or other uncontrolled, severe concurrent infection .
25. Current infection > or equal to Grade 2 (NCI-CTCAE).
26. Any previous or concurrent cancer different to colorectal carcinoma within 5 years before to start the treatment. Subjects with successfully treated, non-invasive cancers, including cervical cancer in situ, basal cell carcinoma will be allowed to participate in the clinical trial. Or those cancer treated with curative intention without disease evidence in the last 5 years at least
27. Known or suspected allergy or hypersensitivity to any component of bevacizumab, cetuximab, irinotecan, or 5-FU/LV.
28. Any medical, psychological, or social condition that may interfere with the subject's participation in the study or evaluation of the study results.
29. Any psychological, familial or geographic situation that interferes in the adequate follow-up and adherence to the study protocol.
30. Women who are pregnant or breast-feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
progression free survival (PFS) | 5 years

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
Response rate (RR) | 5 years
Radical Resection (R0) surgery rate | 5 years
CTC count basal and correlate to PFS, OS, RR | 5 years
Adverse events | 5 years
Correlation of molecular status of bio markers related to the cellular and tumoral reproduction and/or mode of action and clinical anti-tumour activity outcome ( PFS, OS, RR) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Díaz-Rubio, MD-PhD, Study Chair — Hospital San Carlos, Madrid; Enrique Aranda, MD-PhD, Study Chair — Hospital Reina Sofía; Javier Sastre, MD-PhD, Study Chair — Hospital San Carlos, Madrid
Locations (1):
- Spanish Cooperative Group for Digestive Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Valladares-Ayerbes M, Toledano-Fonseca M, Grana B, Jimenez-Fonseca P, Pulido-Cortijo G, Gil S, Sastre J, Salud A, Rivera F, Salgado M, Garcia-Alfonso P, Lopez Lopez R, Guillen-Ponce C, Rodriguez-Ariza A, Vieitez JM, Diaz-Rubio E, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD). Associations of blood RNA biomarkers and circulating tumour cells in patients with previously untreated metastatic colorectal cancer. BMC Cancer. 2025 Apr 21;25(1):743. doi: 10.1186/s12885-025-14098-9. PMID 40259317
- [Derived] Jimenez-Fonseca P, Sastre J, Garcia-Alfonso P, Gomez-Espana MA, Salud A, Gil S, Rivera F, Reina JJ, Quintero G, Valladares-Ayerbes M, Safont MJ, La Casta A, Robles-Diaz L, Garcia-Paredes B, Lopez Lopez R, Guillot M, Gallego J, Alonso-Orduna V, Diaz-Rubio E, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors (TTD). Association of Circulating Tumor Cells and Tumor Molecular Profile With Clinical Outcomes in Patients With Previously Untreated Metastatic Colorectal Cancer: A Pooled Analysis of the Phase III VISNU-1 and Phase II VISNU-2 Randomized Trials. Clin Colorectal Cancer. 2023 Jun;22(2):222-230. doi: 10.1016/j.clcc.2023.02.004. Epub 2023 Feb 21. PMID 36944559
- [Derived] Sastre J, Orden V, Martinez A, Bando I, Balbin M, Bellosillo B, Palanca S, Peligros Gomez MI, Mediero B, Llovet P, Moral VM, Vieitez JM, Garcia-Alfonso P, Calle SG, Ortiz-Morales MJ, Salud A, Quintero G, Lopez C, Diaz-Rubio E, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors (TTD). Association Between Baseline Circulating Tumor Cells, Molecular Tumor Profiling, and Clinical Characteristics in a Large Cohort of Chemo-naive Metastatic Colorectal Cancer Patients Prospectively Collected. Clin Colorectal Cancer. 2020 Sep;19(3):e110-e116. doi: 10.1016/j.clcc.2020.02.014. Epub 2020 Mar 6. PMID 32278676
- See also: Related Info — http://www.ttdgroup.org